CLINICAL TRIAL: NCT01975480
Title: Efficacy of Serotonin-Norepinephrine Reuptake Inhibitor (SNRI) Treatment on Prefrontality in Patients With Generalized Anxiety Disorder (GAD) and Other Comorbidities
Brief Title: Efficacy of SNRI Treatment on Prefrontality in Patients With GAD and Other Comorbities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: START Clinic for Mood and Anxiety Disorders (Other)
Responsible Party: Principal Investigator, Dr. Martin A. Katzman, Principal Investigator, START Clinic for Mood and Anxiety Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS2382578
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Masking Description: Open Label.

ARMS (1):
- Desvenlafaxine (Experimental): At the screening visit those who are eligible will enter a randomized trial with Pristiq (desvenlafaxine) 50 to 100 mg. The study will begin with a single week of Pristiq (desvenlafaxine) 50mg. Subsequently, tablets will be administered in a flexible dose fashion and patients will be followed up weekly (biweekly after week 8) and at the investigators discretion. After the first week the patients' dosage will be increased up to a maximum of 100 mg daily. This dose will remain fixed after 8 weeks of treatment until week 16.
  Interventions: Drug: Desvenlafaxine

INTERVENTIONS:
Drug: Desvenlafaxine
  Other Names: Pristiq

SUMMARY:
This is an open-label flexible-dose pilot study evaluating the efficacy, safety, and tolerability of Pristiq (desvenlafaxine) in outpatient subjects diagnosed with Generalized Anxiety Disorder (GAD) with or without comorbidities that are secondary to the GAD. Primary trial objective is to evaluate the efficacy of Pristiq (desvenlafaxine) SNRI treatment 50 to 100 mg once daily in the treatment of GAD with or without comorbidities. Secondary trial objective is to determine whether or not treatment outcome in GAD is related to changes in cortical prefrontal activity of norepinephrine.

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided signed informed consent.
* Outpatients aged 18-65 (extremes included).
* Patients with a primary diagnosis of GAD according to DSM IV (300.23) criteria (diagnosis to be made using the Mini International Neuropsychiatric Interview; MINI Version 6.0.0). Patients with co-morbid anxiety disorders will be permitted, as long as GAD is judged to be the primary diagnosis.
* Patients who score a HAM-A of ≥ 20 at both Screening and Baseline, and ≥ 10 on the psychic and somatic anxiety factors.
* On the basis of physical examination, medical history, and basic laboratory screening, patient is, in the investigator's opinion, in a suitable condition.
* Willing and able to attend study appointments in the correct time windows.

Exclusion Criteria:

* Any other axis I diagnosis that was a primary disorder in the previous six months.
* Alcohol or drug abuse as defined in the DSM IV (300.23) within the last six months.
* Mania, hypomania as defined in the DSM IV (300.23).
* Any psychotic disorder.
* Eating disorders as defined in the DSM IV (300.23).
* Any cognitive disorder or dementia within 3 months before the baseline visit.
* Clinical interpretation of apparent suicide risk.
* Continuation or commencement of formal psychotherapy.
* Current use of or commencement of antidepressant and anxiolytic medications.
* Failure on no more than 2 antidepressants (either SSRIs or SNRIs to exclude any treatment resistance.
* Patients, who have been on an antidepressant or other anxiolytic prior to the study, will have discontinued it more than two weeks prior to entry into the study. Those who have been on fluoxetine, will have been off of it for at least 5 weeks.
* Patients who have been on a herbal or alternative treatment judged to be potentially anxiolytic or with psychobiological activity (e.g. St. John's Wort, S-adenosylmethionine), will have terminated usage of the agent more than two weeks prior to entering the study.
* Scores on the Hamilton Depression Rating Scale (HAM-D) > 15, at screening visit 1
* Laboratory values at screening or in medical history that may be considered through clinical interpretation to be significant.
* Diseases that could through clinical interpretation interfere with the assessments of safety, tolerability and efficacy.
* Serious illness: Liver or renal insufficiency, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic or metabolic disturbance.
* If female, the subject is pregnant or lactating or intending to become pregnant before, during or within 30 days after participating in this study; or intending to donate ova during such time period.
* The subject has received electroconvulsive therapy, vagal nerve stimulation, or repetitive transcranial magnetic stimulation within 6 months prior to Screening.
* The patient is, in the opinion of the investigator, unlikely to comply with the clinical trial protocol or is unsuitable for any reason.
* Known allergy or intolerance to desvenlafaxine or its excipients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-01; Primary Completion 2020-04-15 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Mean changes in the Hamilton Anxiety Rating Scale from baseline visit to week 16. | 16 weeks

SECONDARY OUTCOMES:
Mean change from baseline to week 16 on the measures of prefrontality including: Frontal System Behavioural Scale and Behaviour Rating Inventory of Executive Function-Adult | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- START Clinic for Mood and Anxiety Disorders, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided